CLINICAL TRIAL: NCT03748134
Title: A Multicenter, Double-Blind, Randomized Phase 3 Clinical Trial Evaluating the Efficacy and Safety of Sintilimab vs. Placebo, in Combination With Chemotherapy, for First-Line Treatment of Unresectable, Locally Advanced, Recurrent, or Metastatic Esophageal Squamous Cell Carcinoma (ORIENT-15)
Brief Title: Sintilimab or Placebo With Chemotherapy in Esophageal Squamous Cell Carcinoma ( ORIENT-15 )
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Collaborators: Fortrea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIBI308A301; 2020-000533-40 (Registry Identifier: EudraCT)
Record Dates: First submitted 2018-11-12; First posted 2018-11-20 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: ESCC; Esophageal Cancer; Esophageal Neoplasms; Esophageal Neoplasms Malignant; Esophageal Squamous Cell Carcinoma; Neoplasms, Squamous Cell; Esophageal Diseases; Carcinoma, Squamous Cell; Gastrointestinal Diseases; Paclitaxel; Cisplatin; Fluorouracil; Antineoplastic Agents; Anti-PD-1; Sintilimab
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms; Neoplasms, Squamous Cell; Esophageal Diseases; Carcinoma, Squamous Cell; Gastrointestinal Diseases | interventions — sintilimab; Cisplatin; Paclitaxel; Fluorouracil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Randomized Part: Experimental: Sintilimab + chemotherapy (Experimental): Sintilimab in combination with investigator's choice of chemotherapy
  TP regimen: Cisplatin + paclitaxel
  or
  CP regimen: Cisplatin + fluorourcil
  Interventions: Biological: Sintilimab; Drug: Cisplatin; Drug: Paclitaxel; Drug: Fluorouracil
- Randomised Part: Active Comparator: Placebo + chemotherapy (Active Comparator): Placebo in combination with investigator's choice of chemotherapy TP regimen: Cisplatin + paclitaxel or CP regimen: Cisplatin + fluorourcil
  Interventions: Drug: Cisplatin; Drug: Paclitaxel; Drug: Fluorouracil; Drug: Placebo
- Open-label part: Sintilimab+ chemotherapy (Experimental): Sintilimab in combination with investigator's choice of chemotherapy TP regimen: Cisplatin + paclitaxel or CP regimen: Cisplatin + fluorourcil
  Interventions: Biological: Sintilimab; Drug: Cisplatin; Drug: Paclitaxel; Drug: Fluorouracil

INTERVENTIONS:
Biological: Sintilimab — For weight <60kg, 3mg/kg IV Q3W day 1, and for weight≥60kg, 200mg IV Q3W day 1
  Arms: Open-label part: Sintilimab+ chemotherapy; Randomized Part: Experimental: Sintilimab + chemotherapy
Drug: Cisplatin — 75mg/m^2 IV Q3W day 1
Drug: Paclitaxel — 87.5 mg/m^2 IV Q3W day 1, day 8 for first cycle and 175mg/m^2 IV Q3W day 1 after first cycle
Drug: Fluorouracil — 800 mg/m^2 IV continuous infusion over 24 hours daily on Days 1-5 Q3W
Drug: Placebo — For weight <60kg, 3mg/kg IV Q3W day 1, and for weight≥60kg, 200mg IV Q3W day 1
  Arms: Randomised Part: Active Comparator: Placebo + chemotherapy

SUMMARY:
This is a randomized, double-blind multi-center, phase III study comparing the efficacy and safety of sintilimab or placebo in combination with chemotherapy as first-line treatment in subjects with unresectable, locally advanced recurrent or metastatic esophageal squamous cell carcinoma.

After the interim analysis conducted by the iDMC, an open-label assignment of experimental arm therapy will continue in regions outside of China, in order to further evaluate the efficacy and safety of sintilimab in combination with chemotherapy in subjects representing the western population with advanced esophageal squamous cell carcinoma

ELIGIBILITY:
Key Inclusion Criteria:

* Histopathologically confirmed unresectable, locally advanced, recurrent or metastatic ESCC (excluding mixed adenosquamous carcinoma and other histological subtypes)
* ECOG PS of 0 or 1
* Subject must be unsuitable for definitive treatment, such as definitive chemoradiotherapy and/or surgery. For subjects who have received (neo)adjuvant or definitive chemotherapy/radiochemotherapy, time from the completion of last treatment to disease recurrence must be > 6 months Could provide archival or fresh tissues for PD-L1 expression analysis with obtainable results
* Have at least one measurable lesion as per RECIST v1.1

Key exclusion Criteria:

* ESCC with endoscopy-confirmed near-complete obstruction requiring interventional therapy
* Post stent implantation in the esophagus or trachea with risk of perforation
* Received systemic treatment for advanced or metastatic ESCC.
* Received a cumulative dose of cisplatin ≥ 300 mg/m2 and the last cisplatin dose was within 12 months of randomization or the first dose of study treatment in the open-label phase.
* High risk of hemorrhage or perforations due to tumor invasion in adjacent organs (aorta or trachea), or have fistula formation.
* Hepatic metastasis > 50% of the total liver volume.
* Received palliative therapy for a local lesion within 2 weeks prior to the first dose.
* Received systemic treatment with Chinese traditional medicines with anti-cancer indications or immunomodulators (including thymosins, interferons, and interleukins) within 2 weeks prior to the first dose of study treatment.
* Received systemic immunosuppressants within 2 weeks prior to randomization, excluding local use of glucocorticoids administered by nasal, inhaled, or other routes, and systemic glucocorticoids at physiological doses (no more than 10 mg/day of prednisone or equivalents), or glucocorticoids to prevent allergies to contrast media.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 746 (Actual)
Dates: Start 2018-12-24 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2023-07-29 (Actual)

PRIMARY OUTCOMES:
OS in overall population | From date of randomization until the date of death from any cause, assessed up to 40 months.
  To compare the overall survival of sintilimab vs. placebo, in combination with chemotherapy, for first-line treatment in subjects with unresectable, locally advanced, recurrent or metastatic esophageal squamous cell carcinoma (ESCC)
OS in PD-L1 positive population | From date of randomization until the date of death from any cause, assessed up to 40 months.
  To compare the OS of sintilimab vs. placebo, in combination with chemotherapy, for first-line treatment in subjects with PD-L1 positive, unresectable, locally advanced, recurrent or metastatic ESCC

SECONDARY OUTCOMES:
ORR in overall population | From date of randomization up to 28 months.
  To compare the objective response rate between the two treatment arms in ITT population
PFS in overall populationsubjects in ITT population | From date of randomization up to 28 months
  To compare the progression-free survival between the two treatment arms in ITT population
DCR in overall population | From date of randomization up to 28 months
  To compare the disease control rate between the two treatment arms in ITT population
DoR in overall population | From date of randomization up to 28 months
  To compare the duration of response between the two treatment arms in ITT population
ORR - PD-L1 positive | From date of randomization up to 28 months
  To compare the objective response rate between the two treatment arms in PD-L1 positive subjects in ITT population
DCR - PD-L1 positive | From date of randomization up to 28 months
  To compare the disease control rate between the two treatment arms in PD-L1 positive subjects in ITT population
DoR - PD-L1 positive | From date of randomization up to 28 months
  To compare the duration of response between the two treatment arms in PD-L1 positive subjects in ITT population
PFS - PD-L1 positive | From date of randomization up to 28 months
  To compare the progression-free survival between the two treatment arms in PD-L1 positive subjects in ITT population

CONTACTS AND LOCATIONS:
Locations (47):
- United States (7):
  - St. Joseph Heritage Healthcare - Virginia K. Crosson Cancer Center, Anaheim, California
  - UC Irvine, Orange, California
  - Rocky Mountain Cancer Centers, LLP, Denver, Colorado
  - IACT Health - John B. Amos Cancer center, Columbus, Georgia
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Texas Oncology, P.A., Austin, Texas
  - Northwest Cancer Specialists, P.C., Vancouver, Washington
- Australia (5):
  - Border Medical Oncology, East Albury, New South Wales
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Austin Hospital, Heidelberg, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - St John of God Subiaco Hospital, Subiaco, Western Australia
- Belgium (5):
  - University Hospital Gent, Ghent, Corneel Heymanslaan 10
  - Universitair Ziekenhuis Leuven, Leuven, Herestraat 49
  - Cliniques Universitaires Saint-Luc Av., Brussels, Hippocrate 10
  - Institut Jules Bordet, Brussels
  - Centre Hospitalier Regional de Verviers, Verviers
- Beijing Cancer Hospital, Beijing, China
- France (12):
  - Hôpital Jean Minjoz, Bettancourt-la-Ferrée
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - CHU Estaing, Clermont-Ferrand
  - Faculte de Medecine, Dijon
  - Universite de Bourgogne - Faculte de Medecine - INSERM U866, Dijon
  - Oscar Lambret Centre, Lille
  - CHU Hôpital de la Timone, Marseille
  - Hôpital Européen Georges Pompidou, Paris
  - CHU de Poitiers, Poitiers
  - Hôpital Charles-Nicolle de Rouen, Rouen
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
- Hungary (2):
  - Országos Onkológiai Intézet, Budapest, Ráth György U. 7-9
  - Jósa András Oktatókórház, Nyíregyháza, Szent István U. 68
- Spain (15):
  - University Hospital Marqués de Valdecilla, Santander, Cantabria
  - Hospital del Mar, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario de Fuenlabrada, Fuenlabrada
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona
  - Hospital Universitari Arnau de Vilanova de Lleida, Lleida
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Clínica Universidad de Navarra, Pamplona
  - Parc Taulí Sabadell Hospital Universitari, Sabadell
  - Complexo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario Virgen Macarena, Seville
  - Consorci Hospital General Universitari de València, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lu Z, Kong L, Wang B, Wang J, Liu L, Shu Y, Yang L, Sun G, Cao G, Ji Y, Cui T, Liu H, Qiu W, Li N, Li G, Luo H, Hou X, Zhang Y, Yue W, Xue L, Liu Z, Pan Y, Gao S, Wang X, Pan Z, Zhang S, Lin G, Xie Y, Gu K, Ren T, Li W, Li T, Wang S, He W, Fan Y, Liang J, Xia B, Zhao L, Wang S, Shen L. Effects of sintilimab plus chemotherapy as first-line treatment on health-related quality of life in patients with advanced esophageal squamous cell carcinoma: results from the randomized phase 3 ORIENT-15 study. EClinicalMedicine. 2024 May 17;72:102623. doi: 10.1016/j.eclinm.2024.102623. eCollection 2024 Jun. PMID 38800802
- [Derived] Zhang Y, Li C, Du K, Pengkhun N, Huang Z, Gong M, Li Y, Liu X, Li L, Wang D, Wang C, Chen F, Li J. Comparative analysis of immune checkpoint inhibitors in first-line treatment of esophageal squamous cell carcinoma: a network meta-analysis. Immunotherapy. 2023 Jul;15(10):737-750. doi: 10.2217/imt-2022-0236. Epub 2023 May 4. PMID 37139963
- [Derived] Lu Z, Wang J, Shu Y, Liu L, Kong L, Yang L, Wang B, Sun G, Ji Y, Cao G, Liu H, Cui T, Li N, Qiu W, Li G, Hou X, Luo H, Xue L, Zhang Y, Yue W, Liu Z, Wang X, Gao S, Pan Y, Galais MP, Zaanan A, Ma Z, Li H, Wang Y, Shen L; ORIENT-15 study group. Sintilimab versus placebo in combination with chemotherapy as first line treatment for locally advanced or metastatic oesophageal squamous cell carcinoma (ORIENT-15): multicentre, randomised, double blind, phase 3 trial. BMJ. 2022 Apr 19;377:e068714. doi: 10.1136/bmj-2021-068714. PMID 35440464